CLINICAL TRIAL: NCT03708588
Title: Chewed Versus Integral Pill of Ticagrelor in All Patients Undergoing Percutaneous Coronary intervention--a Platelet Reactivity and Patient Outcomes Study.
Brief Title: Chewed Versus Integral Pill of Ticagrelor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-078_18-911
Record Dates: First submitted 2018-10-10; First posted 2018-10-17 (Actual); Results first posted 2023-01-18 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2022-11

CONDITIONS: Percutaneous Coronary Intervention
Keywords: Ticagrelor; Stent
MeSH Terms: interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Chewed ticagrelor (Experimental): Drug: Ticagrelor chewed pills. The loading dose will be administered as soon as possible by Catheterization Lab staff after a baseline P2Y12 platelet reaction units (PRU) level is drawn and before the end of the PCI. Patients will be asked to chew, but not swallow, allowing for sublingual absorption. (Loading dose 180mg)
  Interventions: Drug: Ticagrelor
- Active Comparator: Integral pill (Active Comparator): Drug: Ticagrelor integral pills. The loading dose will be administered as soon as possible by Catheterization Lab staff after a baseline P2Y12 platelet reaction units (PRU) level is drawn and before the end of the PCI. Patients will swallow the loading dose followed by 25-50mL (milliliter) of water. (180mg)
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — Chewed
  Other Names: Brilinta; Brilique; Possia
  Arms: Experimental: Chewed ticagrelor
Drug: Ticagrelor — Integral
  Other Names: Brilinta; Brilique; Possia
  Arms: Active Comparator: Integral pill

SUMMARY:
Hypothesis The primary question the investigators propose to answer is whether all patients undergoing percutaneous coronary intervention (PCI) with stent deployment who receive chewed ticagrelor will demonstrate more rapid drug absorption and decreased platelet reactivity as compared to integral pill form 1 hour after drug administration.

DETAILED DESCRIPTION:
Hypothesis The primary question the investigators propose to answer is whether all patients undergoing PCI with stent deployment who receive chewed ticagrelor will demonstrate more rapid drug absorption and decreased platelet reactivity as compared to integral pill form 1 hour after drug administration.

Secondary Hypotheses:

1. Major adverse cardiac and cerebrovascular event (MACCE) rate at 30 days and 1 year.

   1. Death
   2. Repeat myocardial infarction
   3. Need for urgent revascularization
   4. Cerebrovascular accident
2. Rate of stent thrombosis and in-stent stenosis at 30 days and 1 year.
3. Bleeding: Defined as major, minor, or minimal bleeding based on thrombolysis in myocardial infarction (TIMI) criteria.

ELIGIBILITY:
Inclusion Criteria:

• All patients presenting to the cardiac catheterization lab for percutaneous coronary intervention.

Exclusion Criteria:

* Age <18 years or Age >89 years
* Known coagulopathy, bleeding diathesis, or active bleeding
* History of recent gastrointestinal or genitourinary bleed within 2 months
* Known chronic therapy with clopidogrel, prasugrel, or ticagrelor
* Major surgery within last 6 weeks
* History of intracranial bleed or intracranial neoplasm
* Suspected aortic dissection
* Severe hemodynamic instability, cardiogenic shock
* Life expectancy <1 year
* Known severe liver or renal disease
* Known HIV treatment
* Any use of Glycoprotein inhibitors (GP IIb-IIIa) 48-hours before the procedure or any use during the procedure
* Any use of Cangrelor during or after the procedure
* Hemoglobin <10 g/dL, platelet (PLT) <100x10^9/L
* Pregnancy
* Known allergy to study medication

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suhail Allaqaband, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora Health Care, St. Luke's Medical Center, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Chewed Ticagrelor: Drug: Ticagrelor chewed pills. The loading dose will be administered as soon as possible by Catheterization Lab staff after a baseline P2Y12 platelet reaction units (PRU) level is drawn and before the end of the percutaneous coronary intervention (PCI). Patients will be asked to chew, but not swallow, allowing for sublingual absorption. (Loading dose 180mg)
  Ticagrelor: Chewed
- Active Comparator: Integral Pill: Drug: Ticagrelor integral pills. The loading dose will be administered as soon as possible by Catheterization Lab staff after a baseline P2Y12 platelet reaction units (PRU) level is drawn and before the end of the percutaneous coronary intervention (PCI). Patients will swallow the loading dose followed by 25-50mL (milliliters) of water. (180mg)
  Ticagrelor: Integral
Period: Overall Study
Arm/Group | Experimental: Chewed Ticagrelor | Active Comparator: Integral Pill
Started | 55 | 57
Completed | 46 | 48
Not Completed | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Chewed Ticagrelor: Drug: Ticagrelor chewed pills. The loading dose will be administered as soon as possible by Catheterization Lab staff after a baseline PRU level is drawn and before the end of the PCI. Patients will be asked to chew, but not swallow, allowing for sublingual absorption. (Loading dose 180mg)
  Ticagrelor: Chewed
- Active Comparator: Integral Pill: Drug: Ticagrelor integral pills. The loading dose will be administered as soon as possible by Catheterization Lab staff after a baseline PRU level is drawn and before the end of the PCI. Patients will swallow the loading dose followed by 25-50mL of water. (180mg)
  Ticagrelor: Integral
- Total: Total of all reporting groups
Arm/Group | Experimental: Chewed Ticagrelor | Active Comparator: Integral Pill | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (10.1) | 64.5 (9.5) | 65.2 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 33 | 36 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 46 | 48 | 94
Region of Enrollment [Number; unit: participants]
  United States | 46 | 48 | 94
Baseline PRU (P2Y12 platelet reaction units) [Median (Inter-Quartile Range); unit: P2Y12 platelet reaction units] — A blood sample was obtained and sent to the laboratory to register a baseline P2Y12 platelet reaction units (PRU) level prior to the randomized method of taking Ticagrelor.
  P2Y12 platelet reaction units | 242.5 [222 to 284] | 256 [205.5 to 288.5] | 245 [216.8 to 287.3]

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Pharmacodynamics
Description: Platelet function was measured using the VerifyNow P2Y12 Assay (Accumetrics, San Diego, CA). This test is a turbidimetric-based optical detection system that measures ADP (Adenosine diphosphate) - induced platelet agglutination using a proprietary algorithm to report values in PRU.
Time Frame: 1 hour
Measure: Median (Inter-Quartile Range); unit: platelet reaction units
Arm/Group | Experimental: Chewed Ticagrelor | Active Comparator: Integral Pill
Number analyzed (Participants) | 46 | 48
platelet reaction units | 142.5 [31 to 230] | 210 [97.5 to 278.5]

2. Secondary Outcome: Number of Participants With Major Adverse Cardiac and Cerebrovascular Event (MACCE)
Description: Measure events such as: death, repeat myocardial revascularization, cerebrovascular accident, stent thrombosis, in-stent stenosis and bleeding.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Chewed Ticagrelor | Active Comparator: Integral Pill
Number analyzed (Participants) | 46 | 48
Participants | 2 | 0

3. Secondary Outcome: Number of Participants With Major Adverse Cardiac and Cerebrovascular Event (MACCE)
Description: as for outcome 2
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Chewed Ticagrelor | Active Comparator: Integral Pill
Number analyzed (Participants) | 46 | 48
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: Procedure (considered any time during procedure), post procedure (considered time after procedure and up to time of discharge), 30 day follow up, and 1 year follow up
Arm/Group | Experimental: Chewed Ticagrelor | Active Comparator: Integral Pill
All-Cause Mortality (participants affected / at risk) | 2/46 | 1/48
Serious Adverse Events (participants affected / at risk) | 6/46 | 3/48
Other Adverse Events (participants affected / at risk) | 0/46 | 5/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Chewed Ticagrelor (N=46) | Active Comparator: Integral Pill (N=48)
Death - Metastatic brain cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Death by metastatic brain cancer, determined by review of the subjects medical record
Death - Intracerebral hemorrhage (Cardiac disorders) | 1 | 0 — Death - intracerebral hemorrhage, determined by review of the subjects medical record
Death - Undetermined (General disorders) | 1 | 0 — Death - Undetermined, could not be determined by review of the subjects medical record
Inpatient hospitalization or prolongation of existing hospitalization (General disorders) | 4 | 2 — Inpatient hospitalization or prolongation of existing hospitalization, determined by review of the subjects medical record
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Chewed Ticagrelor (N=46) | Active Comparator: Integral Pill (N=48)
Access site complication - Hematoma (Blood and lymphatic system disorders) | 0 | 3 — Access site complication - Hematoma, determined by review of subjects medical record
Urgent revascularization (Surgical and medical procedures) | 0 | 1 — Urgent revascularization, determined by review of subjects medical record
Postural hypertension without syncope (Cardiac disorders) | 0 | 1 — Postural hypertension without syncope, determined by review of subjects medical record

LIMITATIONS AND CAVEATS:
Study limitations include the relatively small sample size, single-center design, and lack of pharmacokinetic confirmation of platelet reactivity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT03708588/Prot_SAP_000.pdf